CLINICAL TRIAL: NCT00310817
Title: A Phase II, Randomized, Observer Blind, Multi-Center, Active Controlled Study to Evaluate the Safety and Immunogenicity of Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Children Aged 12-59 Months.
Brief Title: Safety and Immunogenicity of Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Children Aged 12-59 Months.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: V59P7; EUDRACT NUMBER: 2004-001896-21
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-10

CONDITIONS: Meningococcal Meningitis
Keywords: meningitis; children; vaccine
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- MenACWY-CRM(Ad+) 12 to 35 Months (Experimental): Subjects received one dose of MenACWY-CRM conjugate vaccine with adjuvant (Ad+) on day 1 and second dose at 28 days or at 6 months or at 12 months after the first vaccination.
  Interventions: Biological: MenACWY-CRM conjugate vaccine, adjuvanted
- MenACWY-CRM(Ad-) 12 to 35 Months (Experimental): Subjects received one dose of MenACWY-CRM conjugate vaccine without adjuvant (Ad-) on day 1 and second dose either at 28 days or at 6 months or at 12 months after the first vaccination.
  Interventions: Biological: MenACWY-CRM conjugate vaccine, unadjuvanted
- MenACWY-CRM(Ad-) 36 to 59 Months (Experimental): Subjects received one dose of MenACWY-CRM conjugate vaccine without adjuvant on day 1 and second dose on day 169 or day 337.
  Interventions: Biological: MenACWY-CRM conjugate vaccine, unadjuvanted
- MenACWY-PS (36 to 59 Months) (Active Comparator): Subjects received one dose of MenACWY polysaccharide (PS) vaccine on day 1 and second dose of MenACWY-CRM conjugate vaccine without adjuvant on day 169 or day 337.
  Interventions: Biological: MenACWY polysaccharide vaccine

INTERVENTIONS:
Biological: MenACWY-CRM conjugate vaccine, adjuvanted
  Arms: MenACWY-CRM(Ad+) 12 to 35 Months
Biological: MenACWY polysaccharide vaccine
  Arms: MenACWY-PS (36 to 59 Months)
Biological: MenACWY-CRM conjugate vaccine, unadjuvanted
  Arms: MenACWY-CRM(Ad-) 12 to 35 Months; MenACWY-CRM(Ad-) 36 to 59 Months

SUMMARY:
To compare the functional immune response 28 days after administration of one dose of Men ACWY-CRM conjugate vaccine without adjuvant (MenACWY-CRM(Ad-)) with that of a Men ACWY polysaccharide (PS) vaccine

ELIGIBILITY:
Inclusion Criteria:

* healthy 12-<60 month old children;

Exclusion Criteria:

* subjects who have previously received any meningococcal vaccine
* subjects with any serious acute or chronic progressive disease

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 623 (Actual)
Dates: Start 2005-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Drug Information Services, Study Chair — Novartis
Locations (2):
- University of Tampere Medical School, Tampere, Finland
- Oddz. Neuroinfekcji, Szpital Jana Pawla II, Krakow, Samodzielny ZOZ, Lubartów, Poland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at one center in Finland and in two centers in Poland.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- MenACWY-CRM(Ad+) 12 to 35 Months: Subjects received one dose of MenACWY-CRM(Ad+) vaccine on day 1 and second dose at 28 days or at 6 months or at 12 months after the first vaccination.
- MenACWY-CRM(Ad-) 12 to 35 Months: Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose either at 28 days or at 6 months or at 12 months after the first vaccination.
- MenACWY-CRM(Ad-) 36 to 59 Months: Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose on day 169 or day 337.
- MenACWY-PS (36 to 59 Months): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY conjugate vaccine without adjuvant on day 169 or day 337.
Period: Overall Study
Arm/Group | MenACWY-CRM(Ad+) 12 to 35 Months | MenACWY-CRM(Ad-) 12 to 35 Months | MenACWY-CRM(Ad-) 36 to 59 Months | MenACWY-PS (36 to 59 Months)
Started | 207 | 206 | 128 | 82
Completed | 196 | 198 | 120 | 74
Not Completed | 11 | 8 | 8 | 8
Not completed — AE or Death | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 6 | 7
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Inappropriate Enrollment | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 1
Not completed — Unable to classify | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MenACWY-PS (36 to 59 Months): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(Ad-) vaccine on day 169 or day 337.
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM(Ad+) 12 to 35 Months | MenACWY-CRM(Ad-) 12 to 35 Months | MenACWY-CRM(Ad-) 36 to 59 Months | MenACWY-PS (36 to 59 Months) | Total
Number analyzed (Participants) | 207 | 206 | 128 | 82 | 623
Age, Continuous [Mean (Standard Deviation); unit: Months] | 24.1 (6.4) | 23.7 (6.2) | 45.1 (6.7) | 44.7 (6.4) | 31.0 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 107 | 68 | 44 | 329
  Male | 97 | 99 | 60 | 38 | 294

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Human Complement Serum Bactericidal Activity (hSBA) Titers ≥ 1:4, After One Dose Of Either MenACWY-CRM(Ad-) or MenACWY-PS Vaccine In Subjects 36-59 Months Of Age
Description: Immune response of one dose of MenACWY-CRM(Ad-) compared to that of one dose of MenACWY polysaccharide(MenACWY-PS) vaccine, 28 days after administration to subjects aged 36 to 59 months, as measured by the percentage of subjects with human complement serum bactericidal activity (hSBA) titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 28 days after first vaccination.
Population: Analysis was done on per protocol (PP) dataset -subjects in the modified intention to treat population who received one dose of the study vaccine, and provided an evaluable serum sample at baseline and 28 days after the vaccine dose and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-CRM(Ad-) (36 to 59 Months): Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second vaccination on day 169 or day 337.
- MenACWY-PS (36 to 59 Months): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(Ad-)vaccine on day 169 or day 337.
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 Months) | MenACWY-PS (36 to 59 Months)
Number analyzed (Participants) | 101 | 81
percentages of subjects
  MenA (Baseline; N=101,80) | 2 [0 to 7] | 1 [0.032 to 7]
  MenA (28 days after 1st vaccination; N=101,80) | 75 [66 to 83] | 55 [43 to 66]
  MenC (Baseline; N=99,79) | 14 [8 to 23] | 10 [4 to 19]
  MenC (28 days after 1st vaccination; N=99,79) | 60 [49 to 69] | 52 [40 to 63]
  MenW (Baseline; N=100,81) | 17 [10 to 26] | 19 [11 to 29]
  MenW (28 days after 1st vaccination; N=100,81) | 91 [84 to 96] | 67 [55 to 77]
  MenY (Baseline; N=100,79) | 10 [5 to 18] | 11 [5 to 21]
  MenY (28 days after 1st vaccination; N=100,79) | 77 [68 to 85] | 67 [56 to 77]

2. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After One Dose Of Either MenACWY-CRM(Ad-) or MenACWY-PS Vaccine In Subjects 36-59 Months Of Age
Description: Immune response of one dose of MenACWY-CRM(Ad-) compared to that of a MenACWY-PS vaccine, 28 days after administration to subjects aged 36 to 59 months, as measured by the percentages of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 28 days after first vaccination
Population: Analysis was done on per protocol (PP) dataset, Immunogenicity after one dose of vaccine -subjects in the modified intention to treat population who received one dose of the study vaccine, and provided an evaluable serum sample at baseline and 28 days after the vaccine dose and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 Months) | MenACWY-PS (36 to 59 Months)
Number analyzed (Participants) | 101 | 81
percentages of subjects
  MenA (Baseline) | 2 [0 to 7] | 0 [0 to 5]
  MenA (28 days after 1st vaccination) | 61 [51 to 71] | 39 [28 to 50]
  MenC (Baseline; N=99,79) | 5 [2 to 11] | 8 [3 to 16]
  MenC (28 days after 1st vaccination; N=99,79) | 54 [43 to 64] | 39 [28 to 51]
  MenW (Baseline; N=100,81) | 15 [9 to 24] | 14 [7 to 23]
  MenW (28 days after 1st vaccination; N=100,81) | 84 [75 to 91] | 59 [48 to 70]
  MenY (Baseline; N=100,79) | 7 [3 to 14] | 6 [2 to 14]
  MenY (28 days after 1st vaccination; N=100,79) | 67 [57 to 67] | 57 [45 to 68]

3. Secondary Outcome: hSBA Geometric Mean Titers (GMT) After One Dose Of Either MenACWY-CRM(Ad-) or MenACWY-PS Vaccine In Subjects 36-59 Months Of Age
Description: Immune response of one dose of MenACWY-CRM(Ad-) vaccine compared with that of one dose of MenACWY-PS vaccine, 28 days after administration in subjects 36-59 months of age, as measured by hSBA geometric mean titers (GMTs) against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 28 days after first vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 Months) | MenACWY-PS (36 to 59 Months)
Number analyzed (Participants) | 101 | 81
titers
  MenA (Baseline; N=101,80) | 2.06 [2.02 to 2.1] | 2.03 [1.98 to 2.07]
  MenA (28 days after 1st vaccination; N=101,80) | 15 [11 to 20] | 6.82 [4.89 to 9.53]
  MenC (Baseline; N=99,79) | 2.42 [2.22 to 2.65] | 2.54 [2.3 to 2.8]
  MenC (28 days after 1st vaccination; N=99,79) | 7.12 [5.45 to 9.3] | 7.16 [5.31 to 9.65]
  MenW (Baseline; N=100,81) | 3.05 [2.63 to 3.53] | 3.14 [2.66 to 3.7]
  MenW (28 days after 1st vaccination; N=100,81) | 24 [18 to 31] | 12 [8.68 to 16]
  MenY (Baseline; N=100,79) | 2.42 [2.21 to 2.66] | 2.46 [2.21 to 2.73]
  MenY (28 days after 1st vaccination; N=100,79) | 21 [15 to 29] | 14 [9.99 to 21]

4. Secondary Outcome: hSBA GMTs After One Dose of Either MenACWY-CRM(Ad-) or MenACWY-PS Vaccine In Subjects 36-59 Months Of Age
Description: Persistence of functional immune response at 6 or 12 months following administration of one dose of either MenACWY-CRM(Ad-) or MenACWY-PS vaccine in children aged 36 to 59 months, as measured by hSBA GMTs against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 6 months after first vaccination and 12 months after first vaccination
Population: Analysis was done on PP dataset -subset of subjects in the MITT population for the evaluation of immunogenicity after the 1st dose of either MenACWY Ad+/PS vaccine, provided evaluable serum samples at day 169 day 358 and had no major protocol deviation.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- MenACWY-CRM(Ad-) (36 to 59 M6-): Subjects received two doses of MenACWY-CRM(Ad-) on day 1 and day 169 (6 months after the first vaccination).
- MenACWY-CRM( Ad-) (36 to 59 M12-): Subjects received two doses of MenACWY-CRM(Ad-) on day 1 and day 358 (12 months after the first vaccination).
- MenACWY-PS (36-59 M6PS): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(Ad-) vaccine on day 169 (6 months after first vaccination).
- MenACWY-PS (36-59 M12PS): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(-Ad) vaccine on day 358 (12 months after first vaccination).
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 M6-) | MenACWY-CRM( Ad-) (36 to 59 M12-) | MenACWY-PS (36-59 M6PS) | MenACWY-PS (36-59 M12PS)
Number analyzed (Participants) | 48 | 45 | 32 | 36
titers
  MenA | 2.84 [2.17 to 3.73] | 2.51 [1.9 to 3.32] | 2.96 [2.03 to 4.32] | 2.78 [1.95 to 3.96]
  MenC (N=47,45,32,36) | 5.06 [3.43 to 7.46] | 4.3 [2.89 to 6.39] | 3.33 [2.04 to 5.43] | 3.89 [2.45 to 6.16]
  MenW (N=47,45,32,35) | 22 [14 to 33] | 20 [13 to 30] | 9.98 [5.86 to 17] | 13 [7.76 to 21]
  MenY (N=47,45,32,36) | 11 [7.14 to 18] | 18 [11 to 29] | 6.44 [3.86 to 11] | 5.29 [3.26 to 8.57]

5. Secondary Outcome: Percentage of Subjects With hSBA Titers ≥ 1:4 After One Dose Of Either MenACWY-CRM(Ad-) or MenACWY-PS Vaccine In Subjects 36-59 Months Of Age
Description: Persistence of functional immune response at 6 or 12 months following administration of one dose of either MenACWY-CRM(Ad-) or MenACWY-PS vaccine in children aged 36 to 59 months, as measured by the percentage of hSBA titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 6 months after first vaccination and 12 months after first vaccination
Population: Analysis was done on PP dataset- subjects who received a dose of either MenACWY-CRM(Ad+) or MenACWY(Ad-) vaccine or MenACWY-PS vaccine at either 6 or 12 months from the first vaccination, and provided evaluable serum samples at baseline, at 28 days and 50 days after the first vaccine dose and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-CRM(Ad)- (36 to 59 M6-): Subjects received two doses of MenACWY-CRM(Ad-) on day 1 and day 169 (6 months after the first vaccination).
- MenACWY-CRM(Ad-) (36 to 59 M12-): Subjects received two doses of MenACWY-CRM(Ad-) on day 1 and day 358 (12 months after the first vaccination).
Arm/Group | MenACWY-CRM(Ad)- (36 to 59 M6-) | MenACWY-CRM(Ad-) (36 to 59 M12-) | MenACWY-PS (36-59 M6PS) | MenACWY-PS (36-59 M12PS)
Number analyzed (Participants) | 48 | 45 | 32 | 36
percentages of subjects
  MenA (Day 169) | 23 [12 to 37] | 13 [5 to 27] | 19 [7 to 36] | 14 [5 to 29]
  MenC (Day 169; N=47,45,32,36) | 45 [30 to 60] | 42 [28 to 58] | 28 [14 to 47] | 22 [10 to 39]
  MenW (Day 169; N=47,45,32,36) | 94 [82 to 99] | 84 [71 to 94] | 56 [38 to 74] | 61 [43 to 77]
  MenY (Day 169; N=47,45,32,36) | 70 [55 to 83] | 80 [65 to 90] | 53 [35 to 71] | 42 [26 to 59]

6. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After One Dose Of Either MenACWY -CRM(Ad-) or MenACWY-PS Vaccine In Subjects 36-59 Months Of Age
Description: Persistence of functional immune response at 6 or 12 months following administration of one dose of either MenACWY-CRM(Ad-) or MenACWY-PS vaccine in children aged 36 to 59 months, as measured by the percentage of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 6 months after first vaccination and 12 months after first vaccination
Population: Analysis was done on PP dataset -subjects in the MITT who received a dose of either MenACWY-CRM(Ad+) or MenACWY-CRM(Ad-) or MenACWY-PS vaccine at either 6 or 12 months from the 1st vaccination, and provided evaluable serum samples at baseline, at 28 days and 50 days after the 1st vaccine dose and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 M6-) | MenACWY-CRM( Ad-) (36 to 59 M12-) | MenACWY-PS (36-59 M6PS) | MenACWY-PS (36-59 M12PS)
Number analyzed (Participants) | 48 | 45 | 32 | 36
percentages of subjects
  MenA | 10 [3 to 23] | 9 [2 to 21] | 16 [5 to 33] | 14 [5 to 29]
  MenC (N=47,45) | 32 [19 to 47] | 24 [13 to 40] | 19 [7 to 36] | 19 [8 to 36]
  MenW (N=47,45) | 77 [62 to 88] | 76 [60 to 87] | 53 [35 to 71] | 56 [38 to 72]
  Men Y (N=47,45) | 60 [44 to 74] | 64 [49 to 78] | 38 [21 to 56] | 36 [21 to 54]

7. Secondary Outcome: hSBA GMTs After Second Dose Of MenACWY-CRM(Ad-) Vaccine In Subjects 36-59 Months Of Age
Description: Booster effect of a second dose of MenACWY-CRM(Ad-) vaccine administered either 6 or 12 months after an initial dose of MenACWY-CRM(Ad-) or MenACWY-PS vaccine in children aged 36 to 59 months, as measured 21 days after the booster dose by hSBA GMT against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after second vaccination
Population: Analysis was done on per protocol (PP) dataset, Immunogenicity after one dose of vaccine -subjects in the modified intention to treat population who received two doses of the study vaccine, provided an evaluable serum sample at baseline and 28 days after the second dose and had no major protocol deviation.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- MeMenACWY-PS (36-59 M12PS): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(-Ad) vaccine on day 358 (12 months after first vaccination).
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 M6-) | MenACWY-CRM( Ad-) (36 to 59 M12-) | MenACWY-PS (36-59 M6PS) | MeMenACWY-PS (36-59 M12PS)
Number analyzed (Participants) | 48 | 45 | 32 | 36
titers
  MenA | 51 [35 to 75] | 149 [99 to 222] | 72 [48 to 108] | 116 [79 to 169]
  MenC | 129 [83 to 200] | 472 [301 to 739] | 7.33 [4.22 to 13] | 17 [9.92 to 28]
  MenW | 371 [256 to 535] | 1120 [769 to 1632] | 38 [23 to 64] | 82 [50 to 134]
  MenY | 247 [168 to 364] | 911 [613 to 1353] | 22 [13 to 38] | 24 [14 to 40]

8. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 After Second Dose Of MenACWY-CRM(Ad-) Vaccine In Subjects 36-59 Months Of Age
Description: Booster effect of a second dose of MenACWY-CRM(-Ad) vaccine administered either 6 or 12 months after an initial dose of MenACWY-CRM(Ad-) or MenACWY-PS in children aged 36 to 59 months, as measured 21 days after the booster dose by the percentage of subjects with hSBA titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after second vaccination
Population: Analysis was done on PP dataset- subjects who received a dose of either MenACWY-CRM(Ad+) or MenACWY-CRM(Ad-)vaccine or MenACWY-PS vaccine at either 6 or 12 months from the first vaccination, and provided evaluable serum samples at baseline, at 28 days and 50 days after the first vaccine dose and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-PS (36-59 M6PS): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(Ad-) on day 169 (6 months after first vaccination).
- MenACWY-PS (36-59 M12PS): Subjects received one dose of MenACWY PS vaccine on day 1 and second dose of MenACWY-CRM(Ad-) vaccine on day 358 (12 months after first vaccination).
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 M6-) | MenACWY-CRM(Ad-) (36 to 59 M12-) | MenACWY-PS (36-59 M6PS) | MenACWY-PS (36-59 M12PS)
Number analyzed (Participants) | 48 | 45 | 32 | 36
percentages of subjects
  MenA | 92 [80 to 98] | 98 [88 to 100] | 100 [89 to 100] | 94 [81 to 99]
  MenC (N=47,45) | 100 [92 to 100] | 100 [92 to 100] | 44 [26 to 62] | 56 [38 to 72]
  MenW (N=47,45) | 100 [92 to 100] | 100 [92 to 100] | 97 [84 to 100] | 92 [78 to 98]
  MenY (N=47,45) | 100 [92 to 100] | 100 [92 to 100] | 75 [57 to 89] | 75 [58 to 88]

9. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After Second Dose Of MenACWY-CRM(Ad-) Vaccine In Subjects 36-59 Months Of Age
Description: Booster effect of a second dose of MenACWY-CRM(Ad-) vaccine administered either 6 or 12 months after an initial dose of MenACWY-CRM(Ad-) or MenACWY-PS in children aged 36 to 59 months, as measured 21 days after the booster dose by the percentage of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after the second vaccination
Population: Analysis was done on per protocol (PP) dataset - subjects in the modified intention to treat population who received two doses of the study vaccine, provided an evaluable serum sample at baseline and 28 days after the second dose and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-PS (36-59 M12PS): Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(Ad-) vaccine on day 358 (12 months after first vaccination).
Arm/Group | MenACWY-CRM(Ad-) (36 to 59 M6-) | MenACWY-CRM( Ad-) (36 to 59 M12-) | MenACWY-PS (36-59 M6PS) | MenACWY-PS (36-59 M12PS)
Number analyzed (Participants) | 48 | 45 | 32 | 36
percentages of subjects
  MenA | 90 [77 to 97] | 98 [88 to 100] | 97 [84 to 100] | 94 [81 to 99]
  MenC (N=47,45) | 96 [85 to 99] | 100 [92 to 100] | 34 [19 to 53] | 47 [30 to 65]
  MenW (N=47,45) | 100 [92 to 100] | 100 [92 to 100] | 78 [60 to 91] | 89 [74 to 97]
  MenY (N=47,45) | 100 [92 to 100] | 100 [92 to 100] | 66 [47 to 81] | 58 [41 to 74]

10. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 After One Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Immune response of one dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, 28 days after administration to subjects aged 12 to 35 months, as measured by the percentage of subjects with hSBA titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 28 days after first vaccination.
Population: Analysis was done on per protocol (PP) dataset - subjects in the modified intention to treat population who received one dose of the study vaccine, and provided an evaluable serum sample at baseline and 28 days after the vaccine dose and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-CRM(Ad+) (12 to 35 Months): Subjects received one dose of MenACWY-CRM(Ad+) vaccine on day 1 and second dose at 28 days or at 6 months or at 12 months after the first vaccination.
- MenACWY-CRM(Ad-) (12 to 35 Months): Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose either at 28 days or at 6 months or at 12 months after the first vaccination.
Arm/Group | MenACWY-CRM(Ad+) (12 to 35 Months) | MenACWY-CRM(Ad-) (12 to 35 Months)
Number analyzed (Participants) | 200 | 191
percentages of subjects
  MenA (Baseline) | 0 [0 to 2] | 0 [0 to 2]
  MenA (28 days after 1st vaccination) | 82 [75 to 87] | 70 [63 to 77]
  MenC (Baseline; N=198,190) | 5 [2 to 9] | 1 [0 to 4]
  MenC (28 days after 1st vaccination; N=198,190) | 56 [49 to 63] | 49 [42 to 56]
  MenW (Baseline) | 8 [4 to 12] | 6 [3 to 10]
  MenW (28 days after 1st vaccination) | 82 [76 to 87] | 80 [73 to 85]
  MenY (Baseline; N=199,188) | 5 [2 to 8] | 3 [1 to 7]
  MenY (28 days after 1st vaccination; N=199,188) | 67 [60 to 74] | 67 [60 to 74]

11. Secondary Outcome: hSBA GMT After One Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Immune response of one dose of MenACWY-CRM vaccine with adjuvant or without adjuvant, 28 days after administration to subjects aged 12 to 35 months, as measured by hSBA GMTs against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 28 days after first vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- MenACWY-CRM( Ad-) (12 to 35 Months): Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose either at 28 days or at 6 months or at 12 months after the first vaccination.
Arm/Group | MenACWY-CRM(Ad+) (12 to 35 Months) | MenACWY-CRM( Ad-) (12 to 35 Months)
Number analyzed (Participants) | 200 | 191
titers
  MenA (Baseline) | 2 [1.97 to 2.03] | 2 [1.97 to 2.03]
  MenA (28 days after 1st vaccination) | 18 [15 to 23] | 13 [11 to 16]
  MenC (Baseline; N=198,190) | 2.16 [2.03 to 2.3] | 2.05 [1.92 to 2.18]
  MenC (28 days after 1st vaccination; N=198,190) | 7.43 [6.15 to 8.97] | 5.9 [4.87 to 7.15]
  MenW (Baseline) | 2.38 [2.14 to 2.64] | 2.26 [2.03 to 2.52]
  MenW (28 days after 1st vaccination) | 17 [14 to 21] | 16 [13 to 20]
  MenY (Baseline; N=199,188) | 2.18 [2.04 to 2.34] | 2.12 [1.98 to 2.27]
  MenY (28 days after 1st vaccination; N=199,188) | 12 [9.39 to 15] | 12 [9.54 to 15]

12. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After One Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Immune response of one dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, 28 days after administration to subjects aged 12 to 35 months, as measured by the percentage of subjects with human complement serum bactericidal antibody (hSBA) titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 28 days after first vaccination.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-CRM(Ad+) (12 to 35 Months): Subjects received one dose of MenACWY-CRM(Ad+) vaccine with on day 1 and second dose at 28 days or at 6 months or at 12 months after the first vaccination.
Arm/Group | MenACWY-CRM(Ad+) (12 to 35 Months) | MenACWY-CRM(Ad-) (12 to 35 Months)
Number analyzed (Participants) | 200 | 191
percentages of subjects
  MenA (Baseline) | 0 [0 to 2] | 0 [0 to 2]
  MenA (28 days after 1st vaccination) | 72 [65 to 78] | 61 [53 to 68]
  MenC (Baseline; N=198,190) | 3 [1 to 6] | 1 [0.013 to 3]
  MenC (28 days after 1st vaccination; N=198,190) | 47 [40 to 54] | 36 [29 to 44]
  MenW (Baseline) | 6 [3 to 10] | 4 [1 to 7]
  MenW (28 days after 1st vaccination) | 72 [65 to 78] | 69 [62 to 76]
  MenY (Baseline; N=199,188) | 4 [2 to 8] | 2 [1 to 5]
  MenY (28 days after 1st vaccination; N=199,188) | 60 [53 to 67] | 57 [50 to 64]

13. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 After Second Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Immune response to a second dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, administered 28 days after initial dose to subjects aged 12 to 35 months, as measured 21 days after the second dose by the percentage of subjects with hSBA titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after second vaccination
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-CRM(Ad+) 12-35M1+: Subjects received one dose of MenACWY-CRM(Ad+) vaccine on day 1 and second dose on day 28 (1 month after the first vaccination).
- MenACWY-CRM(Ad-) 12-35M1-: Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose on day 28 (1 month after the first vaccination).
Arm/Group | MenACWY-CRM(Ad+) 12-35M1+ | MenACWY-CRM(Ad-) 12-35M1-
Number analyzed (Participants) | 61 | 48
percentages of subjects
  MenA (N=61,47) | 98 [91 to 100] | 91 [80 to 98]
  MenC | 100 [94 to 100] | 94 [83 to 99]
  MenW | 97 [89 to 100] | 98 [89 to 100]
  MenY (N=61,47) | 97 [89 to 100] | 91 [80 to 98]

14. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After Second Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Immune response to a second dose of either MenACWY-CRM vaccine, with adjuvant or without adjuvant, administered 28 days after the initial dose to subjects aged 12 to 35 months, as measured 21 days after the second dose by the percentage of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after second vaccination
Population: Analysis was done on per protocol dataset - subjects in the Modified Intention to treat population who received the two doses of vaccine correctly, and provided evaluable serum samples at the relevant time points, and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad+) 12-35M1+ | MenACWY-CRM(Ad-) 12-35M1-
Number analyzed (Participants) | 61 | 48
percentages of subjects
  MenA (N=61,47) | 98 [91 to 100] | 85 [72 to 94]
  MenC | 98 [91 to 100] | 90 [77 to 97]
  MenW | 97 [89 to 100] | 90 [77 to 97]
  MenY (N=61,47) | 97 [89 to 100] | 83 [69 to 92]

15. Secondary Outcome: hSBA GMTs After Second Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Immune response to a second dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, administered 28 days after the initial dose to subjects aged 12 to 35 months, as measured 21 days after the second dose by hSBA GMTs against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after second vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- MenACWY-CRM (Ad+) 12-35M1+: Subjects received one dose of MenACWY-CRM(Ad+) vaccine on day 1 and second dose on day 28 (1 month after the first vaccination).
- MenACWY-CRM (Ad-)12-35M1-: Subjects received one dose of MenACWY-CRM(Ad-)vaccine on day 1 and second dose on day 28 (1 month after the first vaccination).
Arm/Group | MenACWY-CRM (Ad+) 12-35M1+ | MenACWY-CRM (Ad-)12-35M1-
Number analyzed (Participants) | 61 | 48
titers
  MenA (N=61,47) | 107 [80 to 143] | 39 [26 to 58]
  MenC | 117 [78 to 174] | 104 [67 to 161]
  MenW | 84 [57 to 122] | 61 [42 to 88]
  MenY (N=61,47) | 74 [50 to 110] | 41 [28 to 60]

16. Secondary Outcome: hSBA GMTs After One Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subject 12-35 Months Of Age
Description: Persistence of immune response at 6 or 12 months following administration of one dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, in subjects aged 12 to 35 months, as measured by hSBA GMTs against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 6 months after first vaccination and 12 months after first vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Groups:
- MenACWY-CRM(Ad+) 12-35M6+: Subjects received one dose of MenACWY-CRM(Ad+) vaccine on day 1 and second dose at 6 months after the first vaccination.
- MenACWY-CRM(Ad+) 12-35M12+: Subjects received one dose of MenACWY-CRM(Ad+) vaccine on day 1 and second dose at 12 months after the first vaccination.
- MenACWY-CRM(Ad-) 12-35M6-: Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose at 6 months after the first vaccination.
- MenACWY-CRM(Ad-) 12-35M12-: Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose at 12 months after the first vaccination.
Arm/Group | MenACWY-CRM(Ad+) 12-35M6+ | MenACWY-CRM(Ad+) 12-35M12+ | MenACWY-CRM(Ad-) 12-35M6- | MenACWY-CRM(Ad-) 12-35M12-
Number analyzed (Participants) | 57 | 56 | 56 | 54
titers
  MenA | 3.54 [2.67 to 4.69] | 2.54 [1.91 to 3.37] | 2.66 [2.07 to 3.42] | 2.41 [1.87 to 3.12]
  MenC | 10 [7.21 to 15] | 4.02 [2.78 to 5.82] | 9.07 [6.35 to 13] | 4.79 [3.33 to 6.88]
  MenW (N=57,54,56,54) | 21 [14 to 31] | 19 [12 to 28] | 14 [9.6 to 21] | 8.19 [5.5 to 12]
  MenY (N=57,55,55,52) | 12 [8.1 to 17] | 8.69 [5.88 to 13] | 10 [6.62 to 16] | 10 [6.39 to 16]

17. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 After One Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Persistence of immune response at 6 or 12 months following administration of one dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, in subjects aged 12 to 35 months, as measured by the percentage of subjects with hSBA titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 6 months after first vaccination and 12 months after first vaccination
Population: Analysis was done on PP dataset -subset of subjects in the MITT population for the evaluation of immunogenicity after the 1st dose of either MenACWY Ad+ / Ad- conjugate vaccine who received a booster dose of either Novartis MenACWY Ad+/ Ad- conjugate vaccine, provided evaluable serum samples at day 169 and 358, had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Groups:
- MenACWY-CRM(Ad-) (12-35M12- ): Subjects received one dose of MenACWY-CRM(Ad-) vaccine on day 1 and second dose at 12 months after the first vaccination.
Arm/Group | MenACWY-CRM(Ad+) 12-35M6+ | MenACWY-CRM(Ad+) 12-35M12+ | MenACWY-CRM(Ad-) 12-35M6- | MenACWY-CRM(Ad-) (12-35M12- )
Number analyzed (Participants) | 57 | 56 | 56 | 54
percentages of subjects
  MenA | 26 [16 to 40] | 14 [6 to 26] | 18 [9 to 30] | 9 [3 to 20]
  MenC | 56 [42 to 69] | 34 [22 to 48] | 63 [49 to 75] | 33 [21 to 47]
  MenW | 82 [70 to 91] | 79 [66 to 88] | 77 [64 to 87] | 54 [40 to 67]
  MenY (N=57,56,55,52) | 65 [51 to 77] | 66 [52 to 78] | 67 [53 to 79] | 56 [41 to 70]

18. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After One Dose Of MenACWY-CRM Vaccine, With or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Persistence of immune response at 6 or 12 months after one dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, in subjects aged 12 to 35 months of age, as measured by the percentage of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 6 months after first vaccination and 12 months after first vaccination
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad+) 12-35M6+ | MenACWY-CRM(Ad+) 12-35M12+ | MenACWY-CRM(Ad-) 12-35M6- | MenACWY-CRM(Ad-) 12-35M12-
Number analyzed (Participants) | 57 | 56 | 56 | 54
percentages of subjects
  MenA | 21 [11 to 34] | 13 [5 to 24] | 11 [4 to 22] | 7 [2 to 18]
  MenC | 51 [37 to 64] | 25 [14 to 38] | 57 [43 to 70] | 26 [15 to 40]
  MenW | 72 [58 to 83] | 73 [60 to 84] | 70 [56 to 81] | 50 [36 to 64]
  MenY (N=57,56,55,52) | 58 [44 to 71] | 50 [36 to 64] | 55 [41 to 68] | 46 [32 to 61]

19. Secondary Outcome: hSBA GMT After Second Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Booster effect of a second dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, administered at 6 or 12 months after an initial dose in children aged 12 to 35 months, as measured 21 days after the booster dose by hSBA GMTs against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after the second vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM(Ad+) 12-35M12+ | MenACWY-CRM(Ad-) 12-35M12- | MenACWY-CRM(Ad+) 12-35M6+ | MenACWY-CRM(Ad-) 12-35M6-
Number analyzed (Participants) | 57 | 56 | 57 | 56
titers
  MenA (N=54,56,57,56) | 168 [116 to 242] | 328 [242 to 445] | 141 [104 to 191] | 66 [46 to 94]
  MenC (N=54,56,56,57) | 575 [381 to 866] | 586 [386 to 889] | 252 [168 to 377] | 297 [197 to 449]
  MenW (N=57,55,57,56) | 1238 [878 to 1745] | 1263 [849 to 1879] | 687 [465 to 1015] | 518 [370 to 726]
  MenY (N=52,56,57,55) | 915 [633 to 1322] | 983 [651 to 1483] | 489 [325 to 735] | 302 [211 to 432]

20. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 After Second Dose Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Booster effect of a second dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, administered at 6 or 12 months after an initial dose in children aged 12 to 35 months, as measured 21 days after the booster dose by the percentage of subjects with hSBA titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after second vaccination
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad+) 12-35M12+ | MenACWY-CRM(Ad-) 12-35M12- | MenACWY-CRM(Ad+) 12-35M6+ | MenACWY-CRM(Ad-) 12-35M6-
Number analyzed (Participants) | 56 | 54 | 57 | 56
percentages of subjects
  MenA | 100 [94 to 100] | 96 [87 to 100] | 100 [94 to 100] | 95 [85 to 99]
  MenC | 98 [90 to 100] | 96 [87 to 100] | 100 [94 to 100] | 100 [94 to 100]
  MenW | 98 [90 to 100] | 100 [93 to 100] | 100 [94 to 100] | 100 [94 to 100]
  MenY (N=56,52,57,55) | 100 [94 to 100] | 100 [93 to 100] | 100 [94 to 100] | 100 [94 to 100]

21. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After Second Dose Of MenACWY-CRM Vaccine, With or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Booster effect of a second dose of MenACWY-CRM vaccine, with adjuvant or without adjuvant, administered either at 6 or 12 months after an initial dose in children aged 12 to 35 months, as measured 21 days after the booster dose by the percentage of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 21 days after second vaccination
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad+) 12-35M12+ | MenACWY-CRM(Ad-) 12-35M12- | MenACWY-CRM(Ad+) 12-35M6+ | MenACWY-CRM(Ad-) 12-35M6-
Number analyzed (Participants) | 56 | 54 | 57 | 56
percentages of subjects
  MenA | 100 [94 to 100] | 96 [87 to 100] | 100 [94 to 100] | 91 [80 to 97]
  MenC | 98 [90 to 100] | 96 [87 to 100] | 100 [94 to 100] | 100 [94 to 100]
  MenW | 98 [90 to 100] | 100 [93 to 100] | 100 [94 to 100] | 100 [94 to 100]
  MenY (N=56,52,57,55) | 100 [94 to 100] | 100 [93 to 100] | 100 [94 to 100] | 100 [94 to 100]

22. Secondary Outcome: hSBA GMTs After Two Doses Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subject 12-35 Months Of Age
Description: Persistence of immune response at 12 months following administration of two doses of MenACWY-CRM vaccine, with adjuvant or without adjuvant, in subjects aged 12 to 35 months, as measured by hSBA GMTs against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 12 months after second vaccination
Population: Analysis was done on PP dataset Immunogenicity of a booster dose - subset of subjects in the MITT population who received a booster dose of either MenACWY Ad+/Ad- conjugate vaccine, and provided evaluable serum samples at day 169, 358 & had no major protocol deviation.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | MenACWY-CRM(Ad+) 12-35M1+ | MenACWY-CRM(Ad-) 12-35M1-
Number analyzed (Participants) | 61 | 49
titers
  MenA (N=61,48) | 5.24 [3.98 to 6.89] | 4.15 [3.16 to 5.45]
  MenC | 13 [8.86 to 18] | 18 [12 to 28]
  MenW (N=61,47) | 29 [20 to 42] | 25 [17 to 37]
  MenY (N=61,48) | 19 [13 to 27] | 19 [12 to 31]

23. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 After Two Doses Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subjects 12-35 Months Of Age
Description: Persistence of immune response, at 12 months following administration of two doses of MenACWY-CRM vaccine, with adjuvant or without adjuvant, in subjects aged 12 to 35 months of age, as measured by the percentage of subjects with hSBA titers ≥ 1:4 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 12 months after second vaccination
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad+) 12-35M1+ | MenACWY-CRM(Ad-) 12-35M1-
Number analyzed (Participants) | 61 | 49
percentages of subjects
  MenA (N=61,48) | 43 [30 to 56] | 29 [17 to 44]
  MenC | 66 [52 to 77] | 73 [59 to 85]
  MenW (N=61,47) | 89 [78 to 95] | 87 [74 to 95]
  MenY | 80 [68 to 89] | 81 [67 to 91]

24. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8 After Two Doses Of MenACWY-CRM Vaccine, With Adjuvant or Without Adjuvant, In Subject 12-35 Months Of Age
Description: Persistence of immune response, at 12 months following administration of two doses of MenACWY-CRM vaccine, with adjuvant or without adjuvant, in subjects aged 12 to 35 months of age, as measured by the percentage of subjects with hSBA titers ≥ 1:8 against N. meningitidis serogroups A, C, W, and Y.
Time Frame: 12 months after second vaccination
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | MenACWY-CRM(Ad+) 12-35M1+ | MenACWY-CRM(Ad-) 12-35M1-
Number analyzed (Participants) | 61 | 49
percentages of subjects
  MenA (N=61,48) | 38 [26 to 51] | 23 [12 to 37]
  MenC | 59 [46 to 71] | 63 [48 to 77]
  MenW (N=61,47) | 87 [76 to 94] | 85 [72 to 94]
  MenY (N=61,48) | 69 [56 to 80] | 71 [56 to 83]

25. Secondary Outcome: Numbers of Subjects 12 to 59 Months of Age Who Reported Solicited Local and Systemic Adverse Events After Any Vaccination
Description: Safety was assessed as the number of subjects 12 to 59 months of age who reported solicited local and systemic adverse events from day 1 up to and including day 7 after the first or second vaccination(s) with MenACWY-CRM vaccine, with adjuvant or without adjuvant or MenACWY-PS vaccine.
Time Frame: From day 1 through day 7 after first or second vaccination(s)
Population: Analysis was done on Safety dataset - all subjects who received at least one dose of vaccine and with some post-baseline safety data.
Measure: Number; unit: Subjects
Groups:
- MenACWY-PS 36 to 59 Months: Subjects received one dose of MenACWY-PS vaccine on day 1 and second dose of MenACWY-CRM(Ad-) vaccine on day 169 or day 337.
Arm/Group | MenACWY-CRM(Ad+) 12 to 35 Months | MenACWY-CRM(Ad-) 12 to 35 Months | MenACWY-CRM(Ad-) 36 to 59 Months | MenACWY-PS 36 to 59 Months
Number analyzed (Participants) | 205 | 206 | 125 | 81
Subjects
  Any Local | 100 | 109 | 70 | 48
  Injection site tenderness | 73 | 79 | 57 | 42
  Injection site erythema | 60 | 63 | 37 | 19
  Injetion site induration | 37 | 38 | 25 | 15
  Any systemic | 98 | 103 | 53 | 26
  Change in Eating Habits | 31 | 46 | 20 | 10
  Irritability | 68 | 74 | 31 | 12
  Vomiting | 17 | 15 | 9 | 2
  Diarrhea | 22 | 24 | 12 | 1
  Fever (≥ 38°C) | 18 | 23 | 10 | 5
  Other | 44 | 38 | 22 | 11
  Analgesic/Antipyretic Med Used | 39 | 35 | 20 | 11

26. Secondary Outcome: Numbers of Subjects 12 to 59 Months Of Age Who Reported Unsolicited Adverse Events and Serious Adverse Events After Any Vaccination
Description: Safety was assessed as the number of subjects 12 to 59 months of age who reported serious adverse events (SAE), AEs necessitating a physician's visit and/or resulting in premature withdrawal from the study, AEs were to be collected between day 7 and the subsequent visit (approximately 1 month later) after the first or second vaccination(s) of MenACWY-CRM vaccine, with or without adjuvant, or MenACWY-PS vaccine. Any SAE were to be collected throughout the study.
Time Frame: 28 days after first vaccination and 21 days after second vaccination
Population: as for outcome 25
Measure: Number; unit: Subjects
Arm/Group | MenACWY-CRM(Ad+) 12 to 35 Months | MenACWY-CRM(Ad-) 12 to 35 Months | MenACWY-CRM(Ad-) 36 to 59 Months | MenACWY-PS 36 to 59 Months
Number analyzed (Participants) | 205 | 206 | 125 | 81
Subjects
  Any AE | 117 | 99 | 64 | 41
  Possibly/probably related AE | 9 | 9 | 3 | 1
  SAE | 13 | 12 | 11 | 9
  AE leading to discontinuation | 3 | 1 | 0 | 0
  Possibly/probably related SAE | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All solicited adverse events (AEs) were collected upto day 7 after each vaccination.
Description: SAEs, AEs necessitating a physician's visit and/or resulting in premature withdrawal from the study AEs were to be collected between day 7 and the subsequent visit (approximately 1 month later) after the first or second vaccination(s) of MenACWY-CRM(Ad+) or MenACWY-CRM(Ad-) or MenACWY-PS vaccine. Any SAE were to be collected throughout the study.
Groups:
- MenACWY-CRM(Ad+) 12 to 35 Months: Subjects received one dose of MenACWY-CRM(Ad+)vaccine on day 1 and second dose at 28 days or at 6 months or at 12 months after the first vaccination.
- MenACWY-CRM(Ad-) 12 to 35 Months: Subjects received one dose of MenACWY-CRM(Ad-)vaccine on day 1 and second dose either at 28 days or at 6 months or at 12 months after the first vaccination.
- MenACWY-CRM(Ad-) 36 to 59 Months: Subjects received one dose of MenACWY-CRM(Ad+) vaccine on day 1 and second dose on day 169 or day 337.
Arm/Group | MenACWY-CRM(Ad+) 12 to 35 Months | MenACWY-CRM(Ad-) 12 to 35 Months | MenACWY-CRM(Ad-) 36 to 59 Months | MenACWY-PS (36 to 59 Months)
Serious Adverse Events (participants affected / at risk) | 13/205 | 12/206 | 11/125 | 9/81
Other Adverse Events (participants affected / at risk) | 155/205 | 158/206 | 97/125 | 58/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM(Ad+) 12 to 35 Months (N=205) | MenACWY-CRM(Ad-) 12 to 35 Months (N=206) | MenACWY-CRM(Ad-) 36 to 59 Months (N=125) | MenACWY-PS (36 to 59 Months) (N=81)
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 2 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 1
Otitis Media (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 6 | 8 | 6 | 6
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Febrile Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Kawasaki's Disease (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM(Ad+) 12 to 35 Months (N=205) | MenACWY-CRM(Ad-) 12 to 35 Months (N=206) | MenACWY-CRM(Ad-) 36 to 59 Months (N=125) | MenACWY-PS (36 to 59 Months) (N=81)
Diarrhoea (Gastrointestinal disorders) | 23 | 25 | 13 | 1
Vomiting (Gastrointestinal disorders) | 17 | 16 | 9 | 2
Injection Site Erythema (General disorders) | 60 | 63 | 37 | 19
Injection Site Induration (General disorders) | 37 | 38 | 25 | 15
Injection Site Pain (General disorders) | 73 | 79 | 57 | 42
Irritability (General disorders) | 68 | 74 | 31 | 12
Pyrexia (General disorders) | 26 | 33 | 15 | 10
Bronchitis (Infections and infestations) | 10 | 11 | 3 | 3
Nasopharyngitis (Infections and infestations) | 11 | 7 | 3 | 2
Otitis Media (Infections and infestations) | 19 | 16 | 9 | 4
Rhinitis (Infections and infestations) | 13 | 7 | 6 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 18 | 19 | 14 | 7
Somnolence (Nervous system disorders) | 36 | 45 | 29 | 12
Eating Disorder (Psychiatric disorders) | 31 | 46 | 20 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 5 | 6 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days